CLINICAL TRIAL: NCT01931007
Title: Use of Autologous Bone Marrow Aspirate Concentrate in Painful Knee Osteoarthritis, A Randomized Placebo Controlled Pilot Study
Brief Title: Use of Autologous Bone Marrow Aspirate Concentrate in Painful Knee Osteoarthritis
Acronym: BMAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shane A. Shapiro, Orthopedic Consultant, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 12-004459
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Bilateral Primary Osteoarthritis of Knee
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Autologous bone marrow concentrate (Experimental): Subjects with symptomatic mild to moderate bilateral knee osteoarthritis will be enrolled in this study. Bone marrow will be aspirated from the patient's iliac crests and the cellular rich portion will be concentrated. Randomly, one knee will be injected with the autologous bone marrow aspirate concentrate. The contralateral knee will be injected with only sterile saline for placebo.
  Interventions: Drug: Autologous Bone Marrow Aspirate Concentrate
- Placebo (Placebo Comparator): Subjects with symptomatic mild to moderate bilateral knee osteoarthritis will be enrolled in this study. Bone marrow will be aspirated from the patient's iliac crests and the cellular rich portion will be concentrated. Randomly, one knee will be injected with the bone marrow concentrate. The contralateral knee will be injected with only sterile saline for placebo.
  Interventions: Drug: Sterile saline

INTERVENTIONS:
Drug: Autologous Bone Marrow Aspirate Concentrate — Autologous Bone marrow aspirate will be concentrated using Magellan Cell Separator and stem cell kit according to the Standard Operating Procedures is to be injected in the treatment knee. 5ml of treatment cells will be combined with 10 ml of previously separated platelet poor bone marrow plasma and used for injection under ultrasound guidance into one of the subject's painful knees.
  Arms: Autologous bone marrow concentrate
Drug: Sterile saline — Bacteriostatic 0.9% sodium chloride, preservative free manufactured by Hospira will be injected into the control knee.
  Arms: Placebo

SUMMARY:
The overall goal of this study is to develop regenerative cell therapy for use in patients with osteoarthritis (OA). The primary objective of this proposal is to conduct a pilot study that assesses the safety and feasibility of using concentrated bone marrow aspirate containing MSC to treat patients with painful knee OA.

DETAILED DESCRIPTION:
Patients with symptomatic mild to moderate bilateral knee osteoarthritis will be candidates for this pilot study. Baseline data includes radiographs, MRI imaging, clinical data on knee pain and analysis of synovial fluid inflammatory markers. Bone marrow will be aspirated from the patient's iliac crests and the cellular rich portion will be concentrated. Randomly, one knee will be injected with the bone marrow concentrate. The contralateral knee will be injected with only sterile saline for placebo. Follow-up analysis of synovial fluid will be at one week and 6 months after injection; clinical data will be obtained at 3, 6 and 12 months and MRI imaging will be performed at 6 months after injection, with repeat radiographs at 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female subjects are both eligible
2. Subjects must be 18 years of age or older
3. Subjects must have bilateral OA and pain in both knees.
4. Osteoarthritis may be primary or secondary. Knees must have Kellgren-Lawrence Grades 1-3.
5. Subjects must have previously tried 6 weeks of one of the following conservative treatments Activity modification, weight loss; physical therapy, anti-inflammatory or injection therapy
6. Patients can provide written informed consent after the nature of the study is fully explained

Exclusion Criteria:

1. Patients with abnormal hematology, serum chemistry, or urinalysis screening laboratory results.
2. Patients taking anti-inflammatory medications (prescription or over-the-counter), including herbal therapies, within 14 days of baseline visit.
3. Patients taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within the 3 months prior to study entry.
4. Patients receiving injections to the treated knee within 2 months prior to study entry.
5. Patients who are pregnant or currently breast-feeding children.
6. Patients with systemic, rheumatic or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis.
7. Patients with ongoing infectious disease, including HIV and hepatitis
8. Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer, or diabetes
9. Patients participating in a study of an experimental drug or medical device within 30 days of study entry.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Reactions to Concentrated Mesenchymal Stem Cells (MSCs) | 1 year
  Occurrence of adverse reactions to concentrated MSCs from bone marrow aspiration injected into knee joints.

SECONDARY OUTCOMES:
Mean Knee Cartilage | baseline, 6 months, 1 year
  Knee cartilage status will be measured prior to injection, at 6 months following injection, and at 12 months following injection. The cartilage will be measured by MRI at baseline and 6 months using MRI and cartilage sequencing techniques, and knee radiographs at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Shapiro, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shapiro SA, Kazmerchak SE, Heckman MG, Zubair AC, O'Connor MI. A Prospective, Single-Blind, Placebo-Controlled Trial of Bone Marrow Aspirate Concentrate for Knee Osteoarthritis. Am J Sports Med. 2017 Jan;45(1):82-90. doi: 10.1177/0363546516662455. Epub 2016 Sep 30. PMID 27566242
- [Derived] Camilleri ET, Gustafson MP, Dudakovic A, Riester SM, Garces CG, Paradise CR, Takai H, Karperien M, Cool S, Sampen HJ, Larson AN, Qu W, Smith J, Dietz AB, van Wijnen AJ. Identification and validation of multiple cell surface markers of clinical-grade adipose-derived mesenchymal stromal cells as novel release criteria for good manufacturing practice-compliant production. Stem Cell Res Ther. 2016 Aug 11;7(1):107. doi: 10.1186/s13287-016-0370-8. PMID 27515308